CLINICAL TRIAL: NCT02030938
Title: SERI® Surgical Scaffold for Soft Tissue Support in Revision Augmentation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofregen Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMA-SERI-13-001
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Subjects Requiring Revision Breast Augmentation Surgery
Keywords: breast implant; revision augmentation; stretch deformity; fold malposition; bottoming out

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SERI® scaffold implanted breasts (Experimental): SERI® Surgical Scaffold is a knitted, multifilament, bioengineered, silk mesh. It is mechanically strong, biocompatible, BIOSILK® purified, and long term bioresorbable. SERI® Surgical Scaffold is a sterile, single use only mesh and is supplied as a 10 x 25 cm sheet. SERI® Surgical Scaffold provides immediate physical and mechanical stabilization of a tissue defect through the strength and porous (scaffold like) construction of its mesh. When long term bioresorption occurs and the patient's own tissue replaces the implanted scaffold over time the mechanical integrity of the repair is maintained.
  SERI® Surgical Scaffold is indicated for use as a transitory scaffold for soft tissue support and repair to reinforce deficiencies where weakness or voids exist that require the addition of material to obtain the desired surgical outcome.
  Interventions: Device: SERI® Surgical Scaffold

INTERVENTIONS:
Device: SERI® Surgical Scaffold — Standard revision augmentation (with or without implant exchange) with the adjunctive use of SERI® Surgical Scaffold placed intra- or extra-capsularly.

SUMMARY:
An evaluation of the clinical performance of SERI® Surgical Scaffold for soft tissue support in subjects undergoing revision augmentation surgery for increased nipple to inframammary fold distance.

DETAILED DESCRIPTION:
This is a single arm prospective study. Approximately 4 investigational sites will enroll and follow subjects who meet the study criteria.The study will span a total of approximately 18 months: an estimated 6 months for recruitment and 12 months for follow up. 50 subjects will be enrolled in the study. It is anticipated that given an average of 1.5 operated breasts per subject enrolled for Revision Augmentation surgery that 75 implantations of SERI® surgical scaffold will occur.

ELIGIBILITY:
Inclusion Criteria:

* Negative nicotine test at screening visit
* Previous augmentation with silicone-filled or saline-filled breast implants requiring Revision Augmentation surgery for increased nipple:inframammary fold distance
* Well vascularized skin flaps that can be approximated without tension

Exclusion Criteria:

* BMI (Body Mass Index) that is ≥ 30 kg/m2
* Active smoker or have smoked within 6 weeks prior to screening visit
* Pregnant or nursing
* Advanced fibrocystic disease considered to be premalignant without accompanying subcutaneous mastectomy
* Carcinoma of the breast
* Previous mastectomy or lumpectomy
* Abscess or infection in the body at the time of enrollment
* Had any disease, including uncontrolled diabetes (e.g., HbAIc > 8%), that is clinically known to impact wound healing ability. For example: collagen-vascular, connective tissue or autoimmune disorders (e.g., Systemic Lupus, Rheumatoid Arthritis, Scleroderma)
* Subjects with diagnosed diabetes must have HbAIc ≤ 8% within 3 months of enrollment
* Showed tissue characteristics that were clinically incompatible with mammaplasty, such as tissue damage resulting from radiation, inadequate tissue, compromised vascularity or ulceration
* Had, or was under treatment for, any condition that may have constituted an unwarranted surgical risk (e.g., unstable cardiac or pulmonary problems)
* History of prior implantation of any surgical scaffold (e.g., synthetic mesh, acellular dermal matrix, or biologic mesh) in the breast
* Implantation of any non-SERI® surgical scaffold (e.g., synthetic mesh, acellular dermal matrix, or biologic mesh) during the study period
* Product contraindications for use of SERI® Surgical Scaffold per the supplied package insert (e.g., hypersensitivity to silk)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Kind, Principal Investigator — Kind Chang Plastic Surgery - California Pacific Medical Center
Locations (5):
- United States (5):
  - Mofid Plastic Surgery, La Jolla, California
  - Kind Chang Plastic Surgery - California Pacific Medical Center, San Francisco, California
  - Somerset Plastic Surgery, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Plastic Surgery Clinic, Mountlake Terrace, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- SERI® Surgical Scaffold Implanted Breasts: SERI® Surgical Scaffold: Standard revision augmentation (with or without implant exchange) with the adjunctive use of SERI® Surgical Scaffold placed intra- or extra-capsularly.
Period: Overall Study
Arm/Group | SERI® Surgical Scaffold Implanted Breasts
Started | 34
Completed | 29
Not Completed | 5
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | SERI® Surgical Scaffold Implanted Breasts
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (13.37)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female - Child-bearing Potential | 22
  Sex: Female - Non Child-bearing Potential | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Reoperation Rate (Per Implanted Breast) for the Presenting Condition at 12 Months.
Description: This refers to the proportion of implanted breasts that will require reoperation for the recurrence of the initial cause of the increase in nipple to inframammary fold distance at the end of the 12-month follow-up period. Reoperation rate outcomes are presented as number of implanted breasts that required a reoperation out of the overall number of units analyzed.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Implanted breasts
Units Other Than Participants: Implanted breasts
Groups:
- Skin Stretch: Subjects who presented with Skin stretch as the initial cause of the increase in N:IMF distance (presenting condition for procedure)
- Fold Malposition: Subjects who presented with Fold Malposition as the initial cause of the increase in N:IMF distance (presenting condition for procedure)
Arm/Group | Skin Stretch | Fold Malposition
Number analyzed (Participants) | 18 | 11
Number analyzed (Implanted breasts) | 34 | 22
Implanted breasts | 0 [0.0 to 10.3] | 0 [0.0 to 15.4]

2. Secondary Outcome: Reoperation Rate (Per Implanted Breast) for Any Cause at 12 Months
Description: This refers to the proportion of implanted breasts that will require reoperation for any cause at the end of the 12 month follow up period. The outcome is presented as the number of implanted breasts that required reoperation from the overall number of units analyzed.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Implanted breasts
Units Other Than Participants: Implanted breasts
Arm/Group | SERI® Surgical Scaffold Implanted Breasts
Number analyzed (Participants) | 29
Number analyzed (Implanted breasts) | 56
Implanted breasts | 1 [0.0 to 9.6]

3. Secondary Outcome: AE Incidence Rates (Per Implanted Breast) at 30 Days
Description: This refers to the AE incidence rate per implanted breast at thirty days. Outcome is reported as the number of adverse events reported for the overall number of units analyzed.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: Adverse events
Units Other Than Participants: Implanted breasts
Arm/Group | SERI® Surgical Scaffold Implanted Breasts
Number analyzed (Participants) | 29
Number analyzed (Implanted breasts) | 56
Adverse events | 1 [0.0 to 9.6]

4. Secondary Outcome: AE Incidence Rates (Per Implanted Breast) at 12 Months
Description: This refers to the AE incidence rate per implanted breast at twelve months. Outcome is reported as the number of adverse events reported for the overall number of units analyzed.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Adverse events
Units Other Than Participants: Implanted breasts
Arm/Group | SERI® Surgical Scaffold Implanted Breasts
Number analyzed (Participants) | 29
Number analyzed (Implanted breasts) | 56
Adverse events | 3 [1.1 to 14.9]

5. Secondary Outcome: Change in Mammometry From Baseline to 12 Months (Per Implanted Breast)
Description: Mammometry is defined as standardized breast measurements. Mammometry was performed by direct measurement (ie with measuring tape) and indirectly through VECTRA imaging.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Implanted breasts
Groups:
- SN:N: Sternal Notch to Nipple distance in cm
- N:IMF: Nipple to Inframammary Fold Distance at rest in cm
Arm/Group | SN:N | N:IMF
Number analyzed (Participants) | 29 | 29
Number analyzed (Implanted breasts) | 54 | 54
cm | -1.42 (7.06) | -1.24 (4.41)

6. Secondary Outcome: Difference in Mean Scores From Baseline to 12 Months Across 4 Scales of the BREAST Q (Per Patient)
Description: The BREAST-Q is a self-administered questionnaire developed at the Memorial Sloan-Kettering Cancer Center and the University of British Columbia. This instrument specifically measured subject satisfaction and health related quality of life (QoL) following different types of breast surgery (reconstruction,augmentation, reduction, and mastectomy only). A subset of 4 scales from the augmentation module (Satisfaction with breasts, Satisfaction with outcome, Psychosocial wellbeing and Sexual wellbeing) were used in this study.
  In accordance with the BREAST-Q manual, subject scores were transformed into linearized measurements on a 0 to 100 scale, using the QScore software which was developed based on the Rasch model. For the transformed scores, a higher score indicated greater satisfaction or higher function.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SERI® Surgical Scaffold Implanted Breasts
Number analyzed (Participants) | 29
units on a scale | 34.8 (24.68)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 12 months
Arm/Group | SERI® Surgical Scaffold Implanted Breasts
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 13/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SERI® Surgical Scaffold Implanted Breasts (N=34)
Breast complication associated with device (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SERI® Surgical Scaffold Implanted Breasts (N=34)
Breast pain (Reproductive system and breast disorders) | 3
Breast mass (Reproductive system and breast disorders) | 2
Breast haematoma (Reproductive system and breast disorders) | 1
Breast swelling (Reproductive system and breast disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Suture rupture (Injury, poisoning and procedural complications) | 1
Physical breast examination abnormal (Investigations) | 1
Physical examination abnormal (Investigations) | 1
Breast complication associated with device (General disorders) | 1
Incision site cellulitis (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Fall (General disorders) | 1
Cutaneous contour deformity (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No